CLINICAL TRIAL: NCT04674592
Title: Biomarkers of Rhabdomyolysis in the Diagnosis of Acute Compartment Syndrome: Study Protocol of a Prospective Multinational, Multicentre Study in Patients With Tibial Fractures.
Brief Title: Biomarkers in the Diagnosis of Acute Compartment Syndrome
Acronym: BioFACTS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Linkoeping (Other)
Collaborators: Medical Research Council of Southeast Sweden (Other Government); Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Jörg Schilcher, Associate professor, University Hospital, Linkoeping
Other Study IDs: BioFACTS
Record Dates: First submitted 2020-12-13; First posted 2020-12-19 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Acute Compartment Syndrome; Tibia Fracture
MeSH Terms: conditions — Tibial Fractures | interventions — Blood Specimen Collection; Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples, muscle biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Tibial fracture: Patients with a traumatic tibial fracture and without acute compartment syndrome.
  Interventions: Other: Blood samples and biopsies
- Tibial fracture complicated by acute compartment syndrome: Patients with a tibial fracture and acute compartment syndrome of fractured leg.
  Interventions: Other: Blood samples and biopsies
- Acute compartment syndrome without fracture: Patients with acute compartment syndrome but without a fracture.
  Interventions: Other: Blood samples and biopsies

INTERVENTIONS:
Other: Blood samples and biopsies — Blood samples for analysis of biomarkers of muscle damage. Muscle biopsies for histological analysis of muscle damage.

SUMMARY:
This prospective multinational, multicentre cohort study aims to investigate the hypothesis that biomarkers of muscle cell damage can predict acute compartment syndrome in patients with tibial fractures.

DETAILED DESCRIPTION:
Patients with a tibial fracture are included. P-myoglobin and P-creatine phosphokinase are analysed at 6-hourly intervals pre- and if applicable, postoperatively after surgical fixation or fasciotomy. Also, blood samples will be collected in 6 hourly intervals if acute compartment syndrome is suspected. An expert panel of senior orthopaedic surgeons will retrospectively assess study data and classify patients who had undergone fasciotomy into those with and without acute compartment syndrome.

Blood samples will also be collected in patients with acute compartment syndrome without tibial fractures, to serve as a positive control group.

ELIGIBILITY:
Tibial fracture group

Inclusion Criteria:

- Traumatic tibial fracture

Exclusion Criteria:

* Malignancy
* Acute myocardial infarction
* Kidney failure (GFR ≤35 ml/min)
* Muscle disease
* Paraplegia/tetraplegia

Non-fracture group

Inclusion Criteria:

- Suspected acute compartment syndrome

Exclusion Criteria:

* Malignancy
* Acute myocardial infarction
* Kidney failure (GFR ≤35 ml/min)
* Muscle disease
* Paraplegia/tetraplegia
* Associated fracture
* Acute vascular event

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a traumatic tibial fracture with or without other concomitant fractures and patients with suspected acute compartment syndrome. The study population is sampled in a consecutive way.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2018-04-05 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Peak levels of P-myoglobin and P-creatine phosphokinase | Up to 5 days
  A series of blood samples will be collected with 6-hourly interval at the following time-points:
  * Admission to hospital: P-myoglobin and P-creatine phosphokinase are collected at 6-hourly intervals for a maximum of 48 hours or until definitive surgical fixation of the fracture is performed (temporary external fixation excluded).
  * Surgical fracture treatment: After surgical intervention (definitive surgical fracture treatment, excluding temporary external fixation), another series of blood samples is collected with 6-hourly interval for 24 hours.
  Acute compartment syndrome: If suspicion of acute compartment syndrome emerges, blood samples will be collected with 6-hourly interval until fasciotomy is performed or the suspicion is written off. After fasciotomy, blood samples will be continued with 6-hourly interval for 24 hours.

SECONDARY OUTCOMES:
MicroRNA | Up to 5 days
  We also collect microRNA specific for muscle damage at the same time intervals and use it as an objective measures of muscle damage.
Histological evidence of muscle damage | At internal fixation and/or fasciotomy
  At surgery (internal fixation or fasciotomy) biopsies are taken from tibialis anterior muscle in some centres for further histological analysis. Two biopsies are taken from the fractured leg, one near the fracture and one at distance, and one biopsy from the uninjured leg (control). Biopsies are frozen within 30 minutes using liquid nitrogen and isopentane and stored in minus 80 degrees Celsius.

CONTACTS AND LOCATIONS:
Overall Officials: Jörg Schilcher, PhD, Principal Investigator — University Hospital, Linkoeping
Locations (1):
- University hospital of Linkoping, Linköping, Sweden

REFERENCES:
- [Derived] Nilsson A, Ibounig T, Lyth J, Alkner B, von Walden F, Fornander L, Ramo L, Schmidt A, Schilcher J. BioFACTS: biomarkers of rhabdomyolysis in the diagnosis of acute compartment syndrome - protocol for a prospective multinational, multicentre study involving patients with tibial fractures. BMJ Open. 2022 May 2;12(5):e059918. doi: 10.1136/bmjopen-2021-059918. PMID 35501102